CLINICAL TRIAL: NCT06592326
Title: A Randomized, Controlled, Open-label, Multicenter Phase 3 Clinical Study of 9MW2821 in Combination With Toripalimab Versus Standard Chemotherapy in First-line Locally Advanced or Metastatic Urothelial Cancer
Brief Title: 9MW2821 in Combination With Toripalimab vs Standard Chemotherapy in Locally Advanced or Metastatic Urothelial Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9MW2821-CP302
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — toripalimab; Gemcitabine; Injections; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9MW2821+Toripalimab (Experimental): 9MW2821+Toripalimab
  Interventions: Drug: 9MW2821; Drug: Toripalimab
- Gemcitabine+Cisplatin/Carboplatin (Active Comparator): Gemcitabine+Cisplatin/Carboplatin
  Interventions: Drug: Gemcitabine; Drug: Cisplatin/Carboplatin

INTERVENTIONS:
Drug: 9MW2821 — 9MW2821, 1.25mg/kg, intravenous (IV) infusion
  Arms: 9MW2821+Toripalimab
Drug: Toripalimab — Toripalimab, 240mg, intravenous (IV) infusion
  Other Names: Toripalimab injection
  Arms: 9MW2821+Toripalimab
Drug: Gemcitabine — Gemcitabine: 1000mg/m2, intravenous (IV) infusion
  Other Names: Gemcitabine Hydrochloride for Injection
  Arms: Gemcitabine+Cisplatin/Carboplatin
Drug: Cisplatin/Carboplatin — Cisplatin: 70mg/m2 or Carboplatin: AUC=4.5/5, intravenous (IV) infusion.
  Other Names: Cisplatin for injection/Carboplatin Injection
  Arms: Gemcitabine+Cisplatin/Carboplatin

SUMMARY:
This is a randomized, controlled, open-label, multicenter phase 3 clinical study to evaluate the efficacy, safety and immunogenicity of 9MW2821 combined with Toripalimab versus standard chemotherapy in first-line locally advanced or metastatic urothelial cancer.

DETAILED DESCRIPTION:
The study is planning to enroll approximately 460 participants with unresectable locally advanced or metastatic urothelial cancer who have not previously received systematic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form approved by IEC.
* Male or female subjects aged 18 to 80 years.
* ECOG status: 0 or 1.
* Histologically confirmed local advanced or metastatic urothelial cancer
* Previously untreated with local advanced or metastatic urothelial cancer
* At least one measurable lesion, according to RECIST V1.1.
* Adequate tumor tissues submitted for test
* Suitable for cisplatin/carboplatin-based chemotherapy assessed by investigator
* Life expectancy for more than 12 weeks.
* Adequate organ functions.
* Proper contraception methods.
* Willingness to follow the study procedures.

Exclusion Criteria:

* History of another malignancy within 3 years.
* History of autoimmune disease requiring systemic treatment within 2 years.
* History of clinically significant cardiac/cerebrovascular diseases or thrombosis within 6 months.
* Major surgery treated within 28 days; Any live vaccines got within 28 days; Radiotherapy or Intravesical therapy treated within 21 days; Traditional Chinese medicine or any potent CYP3A4 inducers/inhibitors taken within 14 days.
* Lots of pleural fluid and ascites, uncontrolled bone pain or spinal compression existed within 14 days; Systemic treatment with active infection within 7 days.
* Previously treated with PD-1, PD-L1, PD-L2, CTLA-4 inhibitors; Previously treated with ADCs which target Nectin-4 or are conjugated with payload MMAE; Organ transplantation or allogeneic hematopoietic stem cell transplantation in the past.
* Clinical significantly toxicity Grade ≥ 2 (except alopecia and pigmentation) related to previous treatment.
* Any situations adding the risk of severe dry eye, active keratitis or corneal ulcer, etc.
* Peripheral neuropathy Grade ≥ 2.
* Any other serious chronic or uncontrolled disease.
* Uncontrolled central nervous system metastases or carcinomatous meningitis.
* Active HBV/HCV/HIV infection, etc.
* Known allergic sensitivity to any of the ingredients of the study drug.
* History of drug abuse or mental illness.
* Other conditions unsuitable into the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
BICR-PFS | up to 50 months
  Progression-free survival, assessed by BICR
OS | up to 50 months
  Overall Survival

SECONDARY OUTCOMES:
ORR | Up to 50 months
  Objective response rate, assessed by BICR or investigator
DCR | Up to 50 months
  Disease control rate, assessed by BICR or investigator
DoR | Up to 50 months
  Duration of response, assessed by BICR or investigator
PFS | Up to 50 months
  Progression-free survival, assessed by investigator
AE/SAE | Up to 50 months
  Adverse event, serious adverse event
Immunogenicity | Up to 50 months
  Anti-Drug Antibody (ADA) of 9MW2821

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang J, Liu R, Wang S, Feng Z, Yang H, Gao S, Li X, Yao X, Chen J, Gong Z, Li Y, Li X, Wang S, Hu C, Liu J, Zhang M, Yuan F, Shi B, Lou H, Zhao P, Qiu F, Guo H, Hu B, Xu D, Huang H, Zhang X, Feng M, Wang X, Li G, Liu D, Chen X, Wang P. Bulumtatug Fuvedotin (BFv, 9MW2821), a next-generation Nectin-4 targeting antibody-drug conjugate, in patients with advanced solid tumors: a first-in-human, open-label, multicenter, phase I/II study. Ann Oncol. 2025 Aug;36(8):934-943. doi: 10.1016/j.annonc.2025.04.009. Epub 2025 Apr 25. PMID 40288679